CLINICAL TRIAL: NCT05999552
Title: The Effect of Eye Exercises Applied on Individuals With Eye Refractive Defects on Visual Function and Quality of Life
Brief Title: The Effect of Eye Exercises in Individuals With Eye Refractive Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Halic University (Other); Bahçeşehir University (Other); Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Emine Nur Demircan, Senior Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Eye Exercises
Record Dates: First submitted 2023-07-29; First posted 2023-08-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Individuals With Eye Refraction Defects
Keywords: Ocular Refraction; Eye; Exercise; Life Quality; Ocular vision
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): any exercise program will not be applied and will only be followed.
- Experimental Group (Experimental): eye exercise program will be applied.
  Interventions: Other: Eye exercises

INTERVENTIONS:
Other: Eye exercises — The treatment will be applied in three sessions a week for eight weeks and each session will be approximately 20 minutes. Individuals will do each exercise shown at home as a home program on other days (days when the physiotherapist does not perform the exercise by video call).
  Arms: Experimental Group

SUMMARY:
According to the World Health Organization's statement published in 2014, 43% of visual impairment is overhauled by uncorrected refractive errors. The change of body and angle of light waves while undergoing changes in the environment due to the temperature difference between the environments is called refraction. The refractive errors found in the eye can be discovered as myopia, astigmatism, hyperopia, and presbyopia. As there are different prevalence methods in eye refractive errors in various publications. According to many studies in the literature, eye exercises in many conditions such as convergence collapse, accommodation dysfunction, movement center of the eye, digital eye strain and dry eye are curative and therapeutic without any control. With eye exercises, blood is applied to the ocular region, the humor is stimulated, the tension of the extraocular muscles is reduced, the coordination between the eye muscles is increased, the eye fatigue and stress are reduced. Depending on the effects of these effects, positive changes are seen on vision tests. Although there is a different view in the literature that includes these eye exercises and their benefits, it has been found to be insufficient in current studies. More work needs to be done in this area so that these results can be stated better and more clearly. With this study, investigators aim to shed light on what can be done in this field by filling these residents in the literature and to examine the visual function and quality of life of eye exercises.

ELIGIBILITY:
Inclusion Criteria:

be between the ages of 18-65, Having any refractive or visual impairment (myopia, hyperopia, astigmatism) by an ophthalmologist, not have other eye problems in addition to these vision defects, to score at least 24 on the Standardized Mini Mental Test.

Exclusion Criteria:

having undergone any eye surgery (including laser operations), have a prosthetic eye have congenital vision loss, have any disease that will affect the eyesight. Individuals meeting these criteria will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Nottingham Health profile | baseline, after 8 weeks
  This questionnaire assesses the perception of health-related quality of life. The total score is between 0-600. A high score is an indication of a bad outcome.
National Institute of Ophthalmology Visual Function Scale | baseline, after 8 weeks
  Used to measure vision-related quality of life in patients with chronic eye disease. Overall scores ranged from 0 to 100, with higher scores indicating better quality of life.
Standardized Mini-Mental Test | baseline
  It is a scale that determines the cognitive level of the participants. It consists of eleven questions and is evaluated over 30 points. 24-30 points are normal, 18-23 points mild dementia, 10-17 points dementia, 10 points and below are compatible with severe dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Calp, PT, MSc, Principal Investigator — Halic University
Locations (1):
- Van bölge hastanesi eğitim ve araştırma hastanesi, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Blindness and visual impairment. [Internet]. World Health Organization, 2014.
- [Background] Convergence Insufficiency Treatment Trial (CITT) Study Group. The convergence insufficiency treatment trial: design, methods, and baseline data. Ophthalmic Epidemiol. 2008 Jan-Feb;15(1):24-36. doi: 10.1080/09286580701772037. PMID 18300086
- [Background] Horwood A, Toor S. Clinical test responses to different orthoptic exercise regimes in typical young adults. Ophthalmic Physiol Opt. 2014 Mar;34(2):250-62. doi: 10.1111/opo.12109. Epub 2014 Jan 29. PMID 24471739
- [Background] Cacho Martinez P, Garcia Munoz A, Ruiz-Cantero MT. Treatment of accommodative and nonstrabismic binocular dysfunctions: a systematic review. Optometry. 2009 Dec;80(12):702-16. doi: 10.1016/j.optm.2009.06.011. PMID 19932444
- [Background] Minoonejad H, Barati AH, Naderifar H, Heidari B, Kazemi AS, Lashay A. Effect of four weeks of ocular-motor exercises on dynamic visual acuity and stability limit of female basketball players. Gait Posture. 2019 Sep;73:286-290. doi: 10.1016/j.gaitpost.2019.06.022. Epub 2019 Jul 16. PMID 31398634
- [Background] Morimoto H, Asai Y, Johnson EG, Lohman EB, Khoo K, Mizutani Y, Mizutani T. Effect of oculo-motor and gaze stability exercises on postural stability and dynamic visual acuity in healthy young adults. Gait Posture. 2011 Apr;33(4):600-3. doi: 10.1016/j.gaitpost.2011.01.016. Epub 2011 Feb 19. PMID 21334899